CLINICAL TRIAL: NCT06788301
Title: The Effects of Virtual Reality and External Cooling and Vibration on Dental Anxiety and Pain During Inferior Alveolar Nerve Block in Children: a Randomized Clinical Trial
Brief Title: Dental Anxiety and Pain During Inferior Alveolar Nerve Block in Children: the Effects of Two Distraction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Arif Bolaca, Assist. Prof. Dr., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022DİŞF003
Record Dates: First submitted 2025-01-06; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Dental Anxiety; Pain; Distraction Methods; Local Anesthesia
Keywords: Dental anxiety; Distraction; Local Anethesia; Pain; Pediatric Dentistry
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (VR eyeglasses) (Experimental): In the VR group, patients wore a VR eyeglasses (Oculus Quest 2, Oculustm Go, Facebook Technologies, Auburn, USA) and watched a previously selected favorite cartoon during the IANB procedure.
  Interventions: Procedure: Inferior Alveolar Nerve Block; Device: VR eyeglasses
- Group II (Buzzy device) (Experimental): In the Buzzy device group, the Buzzy® device (MMJ Labs, Atlanta, GA, USA) was placed extra-orally on the site of IANB (right/left mandibula) during the administration of IANB.
  Interventions: Procedure: Inferior Alveolar Nerve Block; Device: Buzzy device
- Group III (Control) (Other): In the control group, patients received conventional behavior management technique (tell-show-do) during the administration of IANB. Prior to the IANB procedure, the instruments to be used and procedure were explained to the patient in phrases suitable for the patient's cognitive level.
  Interventions: Procedure: Inferior Alveolar Nerve Block

INTERVENTIONS:
Procedure: Inferior Alveolar Nerve Block — local anesthesia administration (inferior alveolar nerve block)
Device: VR eyeglasses — VR eyeglasses was used to distarct patients from dental environment during inferior alveolar nerve block.
  Arms: Group I (VR eyeglasses)
Device: Buzzy device — Buzzy device was used to distarct patients from dental environment during inferior alveolar nerve block.
  Arms: Group II (Buzzy device)

SUMMARY:
Objectives: To compare the effectiveness of virtual reality (VR) and external cooling and vibration distraction techniques on dental anxiety and pain in children during inferior alveolar nerve block (IANB).

Materials and Methods: This randomized controlled parallel arm trial included 120 children aged between 6-12 years old who required IANB. Children were randomly divided following three groups: Group I: VR eyeglasses, Group II: Buzzy® device, and Group 3: Control (conventional behavior management technique). Dental anxiety levels were measured by the pulse rate and oxygen saturation level before, during, and after IANB procedure. Pain perception during IANB procedure was assessed using the Face, Legs, Activity, Cry, Consolability (FLACC) Scale, Wong Baker Faces Scale (WBS), and Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
This study was designed as a three-arm parallel randomized controlled trial to compare the effects of virtual reality (VR) and external cooling and vibration on dental anxiety and pain during inferior alveolar nerve block (IANB) in children aged 6 to 12 years old.

The sample size consisted of 120 children, and the patients were randomly divided following three different groups: Group I: VR eyeglasses group, Group II: Buzzy® device group, and Group III: Control group.

Group I (VR eylasses): In the present study, 3D VR eyeglasses (Oculus Quest 2, Oculus Go, Facebook Technologies, Auburn, USA) were used for VR distraction.

Group II (Buzzy® device): In the present study, the Buzzy® device (MMJ Labs, Atlanta, GA, USA), consisting of a bee-shaped vibrating body and removable wing-shaped cold gel packs, was used for external cooling and vibration application.

Group III (Control): In the present study, group III received conventional behavior management technique (tell-show-do) during the administration of IANB.

Administration of IANB: The oral mucosa was dried with air-water spray and topical anesthetic solution (Vemcaine %10 Lidocaine, VEM Co. Ltd., Istanbul, Turkey) was applied to the dry mucosa with a cotton pellet for 1 minute. The patient was asked to open his/her mouth as wide as possible, and then IANB was administred using 2 ml of 4% articaine with 1:100.000 adrenaline (Ultracaine DS® Forte, Sanofi Health Products Co. Ltd., Istanbul, Turkey) using an automatic aspirated Aspiject® carpule syringe (RØNVIG Dental Mfg. A/S, Daugaard, Denmark) with a 35 mm 27 gauge needle at a rate of 1 ml/minute. In order to ensure standardisation, each patient received the same dosage of local anesthetic and the IANB procedure was provided by the same investigator.

Dental anxiety and pain assessment In order to evaluate physiological changes associated with anxiety, oxygen saturation (SpO2) and pulse rate (PR) values were recorded using pediatric fingertip pulse oximeter (ChoiceMMed, Beijing Choice Electronic Technology Co., Ltd, China) 1 minutes before, during, and 1 minutes after the administration of IANB.

For objective assessment of pain during the IANB procedure, the Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Pain Assessment Scale was used. The FLACC scores were assessed by another investigator not involved in the IANB procedure.

The Wong Baker Face (WBS) and the Visual Analog Scale (VAS), two commonly used and valid pain measurment scale for pediatric patients, were used to assess the self perception of pain. Both scales were explained to the patients, and they were asked to choose the facial expression (for WBS) and the number (for VAS) that best reflected their current level of pain during the IANB procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6-12 years without any systemic disease and physical and/or mental disorders,
* Children whose behavior rating were positive and definitely positive according to the Frankl Behavior Scale (FBS),
* Children with no known allergy to any medication or local anesthetic,
* Children who had mandibular primary/permanent molar requiring dental treatment under an IANB,
* Children with no previous experience of local anesthesia.

Exclusion Criteria:

* Children with systemic disease or neurological behaviour disorders,
* Children whose behavior rating were negative and definitely negative according to the FBS,
* Children with history of allergy to any medication or local anesthetic,
* Children who exhibeted any kind of dento-facial abnormality/syndrome that lead to administration of local anesthesia difficult,
* Children with previous experience of local anesthesia, and non-Turkish speaking

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 1 minutes before, during, and 1 minutes after the administration of inferior alveolar nerve block
  The physiological response of dental anxiety to inferior alveolar nerve block was evaluated by parameters of oxygen saturation value.
Pulse rate | 1 minutes before, during, and 1 minutes after the administration of inferior alveolar nerve block
  The physiological response of dental anxiety to inferior alveolar nerve block was evaluated by parameters of pulse rate value.
Objective pain assessment | During the inferior alveolar nerve block procedure.
  For objective assessment of pain during the inferior alveolar nerve block procedure, the Face, Legs, Activity, Cry, Consolability Behavioral Pain Assessment Scale (0-10) was used. (0: no pain, 1-3: mild pain, 4-6: moderate pain, 7-10: severe pain)
Self perception of pain | Immediately after the inferior alveolar nerve block procedure.
  The Wong Baker Face Scale (0-10) was used to assess the self perception of pain. (0: no pain, 10: severe pain)
Self perception of pain | Immediately after the inferior alveolar nerve block procedure.
  The Visual Analog Scale (0-10) was used to assess the self perception of pain. (0: no pain, 10: severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Arif Bolaca, Dr., Study Director — Pamukkale University Faculty of Dentistry; Aybüke ipek Atik, Dr., Principal Investigator — Pamukkale University Faculty of Dentistry
Locations (1):
- Pamukkale University, Faculty of Dentistry, Department of Pediatric Dentistry, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No